CLINICAL TRIAL: NCT04885153
Title: Effects of Oral Fenofibrate on Retinal Thickness and Macular Volume: Assessments on Retinal Endothelial Vascular Dysfunction, Inflammation, and Angiogenesis in Diabetic Retinopathy With Dyslipidemia
Brief Title: Effects of Oral Fenofibrate on Retinal Thickness and Macular Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Gitalisa Andayani, MD, PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FenofibrateRetinaGitalisa
Record Dates: First submitted 2021-01-21; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Retinopathy; Dyslipidemias; Diabetes Mellitus
Keywords: diabetes mellitus; diabetic retinopathy; dyslipidemia; fenofibrate
MeSH Terms: conditions — Diabetic Retinopathy; Dyslipidemias; Diabetes Mellitus | interventions — Fenofibrate

STUDY DESIGN:
Intervention Model Description: Patients were divided into two groups, which were intervention group (simvastatin+fenofibrate) and control group (simvastatin+placebo).
Who Masked: Care Provider
Masking Description: 200 mg of micronized fenofibrate and placebo (lactic acid) were repackaged into identical capsules and then put inside identical plastic pot by the Pharmacy Unit of Cipto Mangunkusumo Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Subjects who were given simvastatin 10 mg and fenofibrate 200 mg.
  Interventions: Drug: Fenofibrate
- Control Group (Placebo Comparator): Subjects who were given simvastatin 10 mg and placebo (lactic acid) 200 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate — Patients were given simvastatin 10 mg and fenofibrate 200 mg daily for three months and were evaluated monthly.
  Arms: Intervention Group
Drug: Placebo — Patients were given simvastatin 10 mg and placebo (lactic acid) 200 mg daily for three months and were evaluated monthly.
  Arms: Control Group

SUMMARY:
Lipid levels in the blood are proposed to play a role in the progression of diabetic retinopathy. Lipid levels can be controlled with dyslipidemic drugs, such as fenofibrate. Fenofibrate is known to prevent diabetic microvascular complications by decreasing cholesterol and triglyceride levels. This study aims to investigate the effects of oral fenofibrate on central macular thickness (CMT) and macular volume, as well as on specific biomarkers of endothelial dysfunction (eNOS), inflammation (VCAM-1), and angiogenesis (VEGF) in DR individuals with dyslipidemia.

DETAILED DESCRIPTION:
This study was a prospective, double-blind, controlled clinical trial. The study was conducted from 2016 to 2017 at Vitreo-retina Clinic, Department of Ophthalmology, RSCM Kirana. The subjects were non-proliferative diabetic retinopathy (NPDR) patients with dyslipidemia or normal lipid profile with treatment. The outcome measures were central macular thickness (CMT), macular volume, endothelial nitric oxide (eNOS), vascular endothelial growth factor (VEGF), vascular cell adhesion molecule 1 (VCAM-1).

The operational definitions used in our study are as follows:

* Blood glucose control: glucose control status based on HbA1c levels within the last 3 month. Normal values < 7%.
* Dyslipidemia: patient is diagnosed with dyslipidemia if at least one out of four lipid profile parameters is above normal limits (LDL cholesterol ≥ 130, mg/dL, total cholesterol ≥ 200 mg/dL, HDL cholesterol < 40 mg/dL, triglyceride ≥ 150 mg/dL) or normal with treatment.
* Diabetic retinopathy: changes in retinal microvascular based on diabetic retinopathy classification
* Endothelial dysfunction: plasma endothelial nitric oxide (eNOS)
* Inflammation: plasma vascular endothelial growth factor (VEGF)
* Angiogenesis: plasma vascular cell adhesion molecule 1 (VCAM-1).
* Central macular thickness: thickness of fovea centralis based on OCT
* Macular volume: the volume of the retina in the central 6 mm of the macula

Subjects with severe renal failure, allergy towards fenofibrate, pregnant women, and subjects who have undergone laser photocoagulation treatment or intravitreal injection in last 6 months, were excluded. Subjects who did not take medication > 20% of scheduled drug doses were dropped out.

Subjects were allocated into two groups with block randomizations. Sample size calculation revealed a minimum sample size of 18 eyes. Subjects in intervention group received 18 mg of simvastatin and 200 mg of fenofibrate once daily for three months, and subjects in control group received 18 mg of simvastatin and placebo.

All subjects underwent eye examination, fundus photo, and macular spectral-domain optical coherence tomography (SD-OCT), as well as monthly blood and urine laboratory tests. All of the subjects were examined for their uncorrected visual acuity with Snellen chart, intraocular pressure, slitlamp biomicroscopy, and funduscopy through condensed 78 D lens. Fundus photo of both eyes of the subjects were taken before intervention, on every monthly follow-up during intervention, and at the end of study. Fundus photo was done using fundus digital camera (Kowa Medical Equipments, Japan). All fundus photos were read by two vitreo-retina consultants as independent readers. Evaluation of DR degree and the presence of diabetic macula edema (DME) was based on standard of ETDRS severity scale. Inter-reader reliability was also analyzed using Kappa coefficient calculation, which was considered to be acceptable if the value was more than 0.6.

Laboratory tests including HbA1c, triglycerides, total cholesterol, HDL cholesterol and LDL cholesterol, and specific eNOS, VEGF, and serum VCAM-1 biologic markers, were examined at baseline prior to drug administration, and at the end of the study after 3 months. In addition, at the beginning of the study, first, second and third month controls were examined for microalbuminuria, SGOT, SGPT, urine creatinine, blood urea, blood creatinine, and eGFR, to monitor the safety of drug delivery.

Data processing was done using IBM Statistic Program for Social Science (SPSS) version 20. All outcomes were numerical variables, comparison of numerical data between the two groups was performed with unpaired t-test if normal data distribution was fulfilled, otherwise non-parametric Mann Whitney test was used if the data was not normally distributed. To assess the difference between two paired data, Wilcoxon test was used.

ELIGIBILITY:
Inclusion Criteria:

* Adults with type 2 DM
* Confirmed DR (with bio-microscopy examination and fundus photos of both eyes)
* Dyslipidemia or normal lipid profile with treatment
* Sign informed consent

Exclusion Criteria:

* Subjects with severe renal failure
* Subjects with allergy towards fenofibrate
* Pregnant women
* Subjects who have undergone laser photocoagulation treatment or intravitreal injection in last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Central Macular Thickness (CMT) at 3 Months | Evaluated at baseline and monthly for three months
  Thickness of fovea centralis based on OCT
Changes from Baseline Macular Volume at 3 Months | Evaluated at baseline and monthly for three months
  Volume of the retina in the central 6 mm of the macula based on OCT
Changes from Baseline Endothelial Nitric Oxide Synthase (eNOS) at 3 Months | Evaluated at baseline and after three months (by the end of the study)
  Enzyme that produces protective molecule of the blood vessels
Changes from Baseline Vascular Endothelial Growth Factor (VEGF) at 3 Months | Evaluated at baseline and after three months (by the end of the study)
  Signaling protein that promotes angiogenesis
Changes from Baseline Vascular Cell Adhesion Molecule-1 (VCAM -1) at 3 Months | Evaluated at baseline and after three months (by the end of the study)
  Protein that functions for cell adhesion

CONTACTS AND LOCATIONS:
Overall Officials: Gitalisa Andayani, MD, PhD, Principal Investigator — Department of Ophthalmology, Cipto Mangunkusumo Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yau JW, Rogers SL, Kawasaki R, Lamoureux EL, Kowalski JW, Bek T, Chen SJ, Dekker JM, Fletcher A, Grauslund J, Haffner S, Hamman RF, Ikram MK, Kayama T, Klein BE, Klein R, Krishnaiah S, Mayurasakorn K, O'Hare JP, Orchard TJ, Porta M, Rema M, Roy MS, Sharma T, Shaw J, Taylor H, Tielsch JM, Varma R, Wang JJ, Wang N, West S, Xu L, Yasuda M, Zhang X, Mitchell P, Wong TY; Meta-Analysis for Eye Disease (META-EYE) Study Group. Global prevalence and major risk factors of diabetic retinopathy. Diabetes Care. 2012 Mar;35(3):556-64. doi: 10.2337/dc11-1909. Epub 2012 Feb 1. PMID 22301125
- [Background] Landmesser U, Hornig B, Drexler H. Endothelial dysfunction in hypercholesterolemia: mechanisms, pathophysiological importance, and therapeutic interventions. Semin Thromb Hemost. 2000;26(5):529-37. doi: 10.1055/s-2000-13209. PMID 11129409
- [Background] Xu J, Zou MH. Molecular insights and therapeutic targets for diabetic endothelial dysfunction. Circulation. 2009 Sep 29;120(13):1266-86. doi: 10.1161/CIRCULATIONAHA.108.835223. No abstract available. PMID 19786641
- [Background] Koshy J, Koshy JM, Thomas S, Kaur G, Mathew T. Should we start all patients with diabetic retinopathy on fenofibrates? Middle East Afr J Ophthalmol. 2013 Oct-Dec;20(4):309-14. doi: 10.4103/0974-9233.120012. PMID 24339680
- [Background] Keech AC, Mitchell P, Summanen PA, O'Day J, Davis TM, Moffitt MS, Taskinen MR, Simes RJ, Tse D, Williamson E, Merrifield A, Laatikainen LT, d'Emden MC, Crimet DC, O'Connell RL, Colman PG; FIELD study investigators. Effect of fenofibrate on the need for laser treatment for diabetic retinopathy (FIELD study): a randomised controlled trial. Lancet. 2007 Nov 17;370(9600):1687-97. doi: 10.1016/S0140-6736(07)61607-9. Epub 2007 Nov 7. PMID 17988728
- [Background] Noonan JE, Jenkins AJ, Ma JX, Keech AC, Wang JJ, Lamoureux EL. An update on the molecular actions of fenofibrate and its clinical effects on diabetic retinopathy and other microvascular end points in patients with diabetes. Diabetes. 2013 Dec;62(12):3968-75. doi: 10.2337/db13-0800. PMID 24264394
- [Background] Wright AD, Dodson PM. Medical management of diabetic retinopathy: fenofibrate and ACCORD Eye studies. Eye (Lond). 2011 Jul;25(7):843-9. doi: 10.1038/eye.2011.62. Epub 2011 Mar 25. PMID 21436845
- [Background] Massin P, Peto T, Ansquer JC, Aubonnet P, MacuFEN Study Investigators FT. Effects of fenofibric acid on diabetic macular edema: the MacuFen study. Ophthalmic Epidemiol. 2014 Oct;21(5):307-17. doi: 10.3109/09286586.2014.949783. Epub 2014 Aug 18. PMID 25133794
- [Background] Forstermann U, Sessa WC. Nitric oxide synthases: regulation and function. Eur Heart J. 2012 Apr;33(7):829-37, 837a-837d. doi: 10.1093/eurheartj/ehr304. Epub 2011 Sep 1. PMID 21890489
- [Background] Gustavsson C, Agardh CD, Zetterqvist AV, Nilsson J, Agardh E, Gomez MF. Vascular cellular adhesion molecule-1 (VCAM-1) expression in mice retinal vessels is affected by both hyperglycemia and hyperlipidemia. PLoS One. 2010 Sep 13;5(9):e12699. doi: 10.1371/journal.pone.0012699. PMID 20856927
- [Background] Hoeben A, Landuyt B, Highley MS, Wildiers H, Van Oosterom AT, De Bruijn EA. Vascular endothelial growth factor and angiogenesis. Pharmacol Rev. 2004 Dec;56(4):549-80. doi: 10.1124/pr.56.4.3. PMID 15602010
- [Background] Saxena S, Khatri M, Nadri G, Ankita. Pathogenic Mechanisms for Outer Retinal Layer Changes in Diabetic Retinopathy. Ann Diabetes Metab Disord Contr. 2017; 1:113.